CLINICAL TRIAL: NCT06476678
Title: Prospective Multicenter Trial Evaluating the Efficacy and Feasibility of a Novel Bipolar Radiofrequency Ablation Knife in Esophageal Endoscopic Submucosal Dissection
Brief Title: Novel Bipolar Radiofrequency Ablation Knife in Esophageal Lesions
Status: Recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: Creo Medical Limited (Industry)
Responsible Party: Principal Investigator, Salmaan Azam Jawaid, MD, Principal Investigator, Baylor College of Medicine
Other Study IDs: H-55206
Record Dates: First submitted 2024-06-21; First posted 2024-06-26 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Esophageal Neoplasm; Esophageal Polyp; Endoscopic Submucosal Dissection; Bipolar Electrocautery
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Treatment arm: Patients who were deemed eligible and signed the consent will undergo the removal of their esophageal precancerous lesion utilizing the novel bipolar knife during their endoscopic submucosal dissection (ESD).
  Interventions: Device: Speedboat™ Ultraslim

INTERVENTIONS:
Device: Speedboat™ Ultraslim — Use of Speedboat™ Ultraslim for performing endoscopic submucosal dissection of esophageal lesions.

SUMMARY:
Both Baylor St Luke's Medical Center and Mayo Scottsdale are considered endoscopic submucosal dissection (ESD) centers of excellence. The investigators at Baylor College of Medicine have previously reported our Esophageal ESD experience using the monopolar current knife. Moreover, the research team have previously reported on the clinical efficacy of the bipolar RFA knife during per-oral endoscopic myotomy (POEM) and colonic ESD. The goal of our study is to prospectively evaluate the efficacy, safety and feasibility of Esophageal ESD using a novel Bipolar-Current ESD device.

DETAILED DESCRIPTION:
Endoscopic submucosal dissection (ESD) is a novel technique for the removal of esophageal lesions or polyps with high-risk features. ESD is minimally invasive and allows the removal of esophageal polyps without resorting to morbid surgery. The process of ESD includes marking the lesions selected for removal, followed by submucosal injection of a lifting agent, then circumferential incisions using a specialized knife followed by submucosal dissection of the entire lesion.

Traditionally, knifes utilizing monopolar current were the preferred tools for endoscopic submucosal dissection. These knifes allow accurate dissection and excellent hemostasis. However, due to monopolar current generated heat, post coagulation syndrome can be seen in up to 8 to 40 % of patients. Post coagulation syndrome present with pain, fever and leukocytosis and requires supportive treatment with IV fluid and antibiotics. In addition, for large esophageal lesions, stricturing can occur after resection due to significant scar formation resulting from the tissue healing response to electrocautery. Almost all patients with >60% of the esophageal circumference removed via monopolar knives, will develop an esophageal stricture at some point. These patients require serial esophageal dilations, and although easily managed, its development can be quite troublesome to the patient. Nevertheless, ESD is still the preferred modality for removal of these lesions since it avoids the need for morbid surgery.

Recently, a novel Bipolar RFA knife was FDA approved for endoscopic submucosal dissection. The low voltage bipolar system allows for precise cutting of submucosa and muscle using substantially less energy, thereby limiting inadvertent remote thermal effects. Additionally, it allows aggressive coagulation of vessels without dissipation of large amounts of energy, thereby allowing more targeted therapy. Moreover, with the addition of an integrated injection needle, the knife now allows injection, safe cutting and coagulation in one device, potentially supporting more efficient dissection. Ultimately, due to less thermal effect on surrounding tissue, the bipolar knife may allow for removal of large esophageal lesions without causing major esophageal stricturing.

ELIGIBILITY:
Inclusion Criteria:

* Patient is >18 years of age
* Patient can provide informed consent
* Patient is referred for resection of precancerous lesions meeting the following criteria:

  * Mucosal based polyp
  * Located gastroesophageal junction (GEJ) or proximal to GEJ
  * No previous endoscopic resection attempted (EMR or ESD)

Exclusion Criteria:

* Patients with International Normalized Ratio (INR) >1.5 or Platelets <50,000
* Lesions extending past GEJ
* Subepithelial lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing intended ESD of precancerous lesions will be screened by study coordinators for preliminary eligibility and those who meet the inclusion criteria will be approach individually for further discussion about the study and obtaining informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Technical success | Day 1 (procedure day)
  Defined as the ability to perform the entire dissection (procedure) with the novel bipolar knife

SECONDARY OUTCOMES:
Speed of Endoscopic Submucosal Dissection | During Procedure
  The speed of endoscopic submucosal dissection as calculated by cm^2/hour
Number of instruments used | During Procedure
  Logging the variable equipment utilized during the procedure
Rate of muscle injury score | During Procedure
  As calculated by the Sydney Classification of Deep Mural Injury ranging from Type 0 - Type V with Type V as the most severe score.
Rate of post-electrocautery syndrome | 24 hours, 2 weeks, and 4 weeks
  Define as post-procedure abdominal pain, fevers, leukocytosis
Change in post-procedural pain score | 24 hours, 2 weeks, and 4 weeks
  As calculated by the visual analog pain scale to measure patient pain ranging from 0-10 with 10 being the most pain.
Rate of esophageal stricturing | Assessed at any follow-up post-procedure endoscopies up to 6 months
  Calculated by number of documented occurrences post-procedure for subjects
Degree of scar formation | Assessed at any follow-up post-procedure endoscopies up to 6 months
  Scar formation that occurs in response to electrocautery
Cost of dissection | During Procedure
  As calculated upon review of devices used during dissection procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States